CLINICAL TRIAL: NCT03203590
Title: Oral Navelbine Carboplatin Versus Gefitinib Neoadjuvant Therapy for Resectable EGFR Mutation Positive Stage Ⅱ-ⅢA NSCLC, Prospective, Randomized, Multicenter, Phase Ⅲ Clinical Trial
Brief Title: Clinical Trial of Neoadjuvant Targeted Treatment to NSCLC Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shenzhen People's Hospital (Other); Dongguan People's Hospital (Other Government); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Maoming Affiliated Hospital of Southern Medical University (Unknown)
Responsible Party: Principal Investigator, Guowei Ma, Professor,Chief Physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3939366
Record Dates: First submitted 2017-06-21; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: 2-year Disease-Free Survival
MeSH Terms: interventions — Vinorelbine; Carboplatin; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Navelbine + Carboplatin (Active Comparator): Neoadjuvant therapy Patients with EGFR mutation will be recruited and treated with Navelbine + Carboplatin.
  Interventions: Drug: Oral Navelbine + Carboplatin
- Gefitinib (Experimental): Neoadjuvant therapy Patients with EGFR mutation will be recruited and treated with gefitinib.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Oral Navelbine + Carboplatin — The patient will be given Navelbine 60 mg/m2, p.o. day 1 and 8 of every cycle (21 days) plus carboplatin AUC 5, i.v. day 1 of every cycle.After 2 cycle we will evaluate their clinical response.Then operable patients will have surgery.
  Other Names: Vinorelbine; Carboplat
  Arms: Oral Navelbine + Carboplatin
Drug: Gefitinib — The patient will be given Gefitinib 250mg,p.o.,q.d. for 8 weeks.After 8 weeks we evaluate their clinical response.Then operable patients will have surgery.
  Other Names: Iressa
  Arms: Gefitinib

SUMMARY:
The purpose of this study is to evaluate the efficiency and safety of Gefitinib Neoadjuvant Therapy and Oral Navelbine Carboplatin Neoadjuvant Therapy for Resectable Stage Ⅱ-ⅢA NSCLC patients with EGFR mutation.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer mortality in men and women in the world. LACE meta analysis shows that the 5-year survival rate of post-operation chemotherapy group rose by 5.4%, therefore, adjuvant chemotherapy has been the main treatment after surgery according to National Comprehensive Cancer Network (NCCN) Guideline. But patients have poor compliance due to physical condition after surgery. Compared with adjuvant chemotherapy, neoadjuvant therapy has better patient compliance and tolerance.Targeted therapy, with milder side effect compared with chemotherapy, may be a promising choice to treat NSCLC previously. But to date, there is no enough evidence to support the efficacy and safety of neoadjuvant targeted therapy in patients with EGFR mutation.The purpose of this study is to evaluate the efficiency and safety of Gefitinib Neoadjuvant Therapy vs Oral Navelbine Carboplatin Neoadjuvant Therapy for Resectable NSCLC patients harboring EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of non small cell lung cancer, Stage Ⅱ-ⅢA before treatment
* EGFR Gene mutated
* ECOG 0-1
* liver, kidney and bone marrow are functional healthy，WBC>4.0×109/L，PLT>100×109/L Hb>10g/dL;Cr<1.8mg/dL，bilirubin<1.5mg/dL，GPT<1.5 upper limit of normal
* No vital systems dysfunction or malnutrition
* No other malignant diseases in 5 years（except non melanoma or Cervical carcinoma in situ）
* Have never accepted radiation therapy、overall chemotherapy or biotherapy
* Know the whole protocol，Voluntary participate and sign a consent form

Exclusion Criteria:

* Tumor has violated the surrounding tissue organs（T4）
* Preoperative have evidence of distant metastasis including the contralateral mediastinal lymph nodes
* Arrhythmia need anti-arrhythmic treatment（except for β-blockers or digoxin），Symptomatic coronary artery disease and myocardial ischemia (myocardial infarction) in the past 6 months or more than NYHA class II congestive heart failure
* Adverse drug control severe hypertension
* Moderate to severe proteinuria
* History of HIV infection or activity of chronic hepatitis b or hepatitis c, or other active clinical severe infection
* Cachexy,organ function decompensation
* History of chest radiotherapy
* Not fully control the eye inflammation
* Epilepsy patients needed treatment（such as Steroids or antiepileptic cure）
* Interstitial pneumonia
* Drug abuse and medical, psychological or social conditions may interfere with the patients involved in the research or have an impact on the results of evaluation
* Known or suspected to study drug allergy or to give any drug allergies associated with this test
* Any unstable situation or may endanger the patient safety and compliance
* Fertility and pregnancy or lactation women, and have not been sufficient precautions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
2-year disease free survival | 2 years

SECONDARY OUTCOMES:
Objective response rate | 1 week before surgery
Pathologic complete response | Within 1 month after surgery
Side effects | 1 week before surgery
Standard uptake value | 1 week before surgery
Tumor reduction rate | Within 1 month after surgery
Mediastinal lymph nodes clearance | Within 1 month after surgery
Postoperative complications | Within 1 month after discharge
R0 resection rate | Within 1 month after surgery
Postoperative mortality rate | Within 1 month after discharge
5-year overall survival | 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guowei Ma, MD, Principal Investigator — Sun Yat-sen University
Locations (5):
- China (5):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Maoming Affiliated Hospital of Southern Medical University, Maoming, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: Yes